CLINICAL TRIAL: NCT07218510
Title: A Phase 2 Study of Venetoclax + Obinutuzumab Followed by Epcoritamab in Previously Untreated Chronic Lymphocytic Leukemia/ Small Lymphocytic Lymphoma (LonGEVity)
Brief Title: Venetoclax and Obinutuzumab Followed by Epcoritamab for the Treatment of Untreated Chronic Lymphocytic Leukemia and Small Lymphocytic Lymphoma, LonGEVity Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24230; NCI-2025-07205 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24230 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Specimen Handling; Biopsy; Magnetic Resonance Spectroscopy; obinutuzumab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (obinutuzumab, venetoclax, epcoritamab) (Experimental): Patients receive obinutuzumab IV on days 1, 2, 8 and 15 of cycle 1 and on day 1 of cycles 2-6, venetoclax PO QD on days 22-28 of cycle 1 and on days 1-28 of cycles thereafter, as well as epcoritamab SC on days 1, 8, 15, and 22 of cycles 7-9 and on day 1 of cycles thereafter. Cycles repeat every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. After completion of 12 cycles, patients who are MRD positive and have CR, PR, or SD continue receiving epcoritamab SC on day 1 of each cycle. Cycles of epcoritamab repeat every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. All patients also undergo blood sample collection and CT or MRI throughout the study. Additionally, patients may undergo bone marrow aspiration and biopsy throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Other: Electronic Health Record Review; Biological: Epcoritamab; Procedure: Magnetic Resonance Imaging; Biological: Obinutuzumab; Drug: Venetoclax

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration and biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Other: Electronic Health Record Review — Ancillary studies
Biological: Epcoritamab — Given SC
  Other Names: Anti-CD20/CD3 Bispecific Antibody GEN3013; DuoBody-CD3xCD20; Epcoritamab-bysp; Epkinly; GEN 3013; GEN-3013; GEN3013; Tepkinly
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Obinutuzumab — Given IV
  Other Names: Anti-CD20 Monoclonal Antibody R7159; GA 101; GA-101; GA101; Gazyva; huMAB(CD20); R 7159; R-7159; R7159; RO 5072759; RO-5072759; RO5072759
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial tests the effect of venetoclax and obinutuzumab followed by epcoritamab in treating patients with chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) that have not previously received treatment. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Obinutuzumab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. A monoclonal antibody is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). Epcoritamab, a bispecific monoclonal antibody, binds to a protein called CD3, which is found on T cells (a type of white blood cell). It also binds to a protein called CD20, which is found on B cells (another type of white blood cell) and some lymphoma cells. This may help the immune system kill cancer cells. The combination of venetoclax and obinutuzumab is a standard treatment for CLL/SLL and has been found to be safe and effective. Adding epcoritamab to standard treatment with venetoclax and obinutuzumab may lead to deeper and longer-lasting responses in patients with untreated CLL/SLL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the efficacy of venetoclax and obinutuzumab followed by venetoclax and epcoritamab in patients with newly diagnosed CLL/SLL, as assessed by the minimal residual disease (MRD)-negative complete response (CR) rate at 12 cycles of therapy.

SECONDARY OBJECTIVES:

I. Evaluate the safety and tolerability of venetoclax and obinutuzumab followed by venetoclax and epcoritamab in patients with newly diagnosed CLL/SLL.

II. Evaluate the overall response rate (ORR), progression-free survival (PFS), duration of response (DOR) and overall survival (OS) in patients with newly diagnosed CLL/SLL who received venetoclax and obinutuzumab followed by venetoclax and epcoritamab.

EXPLORATORY OBJECTIVES:

I. Examine T cell and natural killer (NK) cell immune function in patients with newly diagnosed CLL/SLL treated with venetoclax and obinutuzumab followed by venetoclax and epcoritamab.

II. Examine the association between established biomarkers (chromosomal abnormalities, immunoglobulin heavy chain [IGHV] mutational status, TP53 mutational status) and clinical outcomes (ORR, PFS).

OUTLINE:

Patients receive obinutuzumab intravenously (IV) on days 1, 2, 8 and 15 of cycle 1 and on day 1 of cycles 2-6, venetoclax orally (PO) once daily (QD) on days 22-28 of cycle 1 and on days 1-28 of cycles thereafter, as well as epcoritamab subcutaneously (SC) on days 1, 8, 15, and 22 of cycles 7-9 and on day 1 of cycles thereafter. Cycles repeat every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. After completion of 12 cycles, patients who are MRD positive and have CR, partial response (PR), or stable disease (SD) continue receiving epcoritamab SC on day 1 of each cycle. Cycles of epcoritamab repeat every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity.

All patients also undergo blood sample collection and computed tomography (CT) or magnetic resonance imaging (MRI) throughout the study. Additionally, patients may undergo bone marrow aspiration and biopsy throughout the study.

After completion of study treatment, patients are followed up at 30 and 60 days, then every 6 months (for patients who have not experienced disease progression) and 12 months (after disease progression) for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Histologically confirmed or flow cytometry confirmed diagnosis of B-CLL/SLL as documented by medical records and with histology based on criteria established by the World Health Organization (WHO)
* No prior treatment for CLL/SLL, except steroids and/or rituximab to treat autoimmune complications
* Evidence of CD20 positivity
* Active disease meeting criteria for requiring treatment per the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018 guidelines

  * A minimum of any one of the following constitutional symptoms:

    * Unintentional weight loss > 10% within the previous 6 months prior to screening
    * Extreme fatigue (unable to work or perform usual activities)
    * Fevers of greater than 100.5°F for ≥ 2 weeks without evidence of infection
    * Night sweats without evidence of infection
  * Evidence of progressive marrow failure as manifested by the development of, or worsening of anemia or thrombocytopenia
  * Massive (i.e., > 6 cm below the left costal margin), progressive or symptomatic splenomegaly
  * Massive nodes or clusters (i.e., > 10 cm in longest diameter) or progressive lymphadenopathy
  * Progressive lymphocytosis with an increase of > 50% over a 2-month period, or an anticipated doubling time of less than 6 months
  * Autoimmune anemia or thrombocytopenia that is poorly responsive to corticosteroids
  * Symptomatic or functional extranodal involvement (e.g., skin, kidney, lung, spine)
* Participant must be able to swallow tablets or capsules. A participant with any gastrointestinal disease that would impair ability to swallow, retain, or absorb drug is not eligible
* Without bone marrow involvement: Absolute neutrophil count (ANC) ≥ 1,000/mm^3

  * NOTE: Growth factor is not permitted within 14 days of ANC assessment unless cytopenia is secondary to disease involvement.
* With bone marrow involvement: ANC ≥ 500/mm^3

  * NOTE: Growth factor is not permitted within 14 days of ANC assessment unless cytopenia is secondary to disease involvement.
* Without bone marrow involvement: Platelets ≥ 50,000/mm^3

  * NOTE: independent of transfusion support, with no active bleeding
* With bone marrow involvement: Platelets ≥ 30,000/mm^3

  * NOTE: independent of transfusion support, with no active bleeding
* Direct bilirubin ≤ 2 x upper limit of normal (ULN) (unless has Gilbert's disease or compensated hemolysis directly attributable to CLL)
* Aspartate aminotransferase (AST) ≤ 2.5 x ULN
* Alanine aminotransferase (ALT) ≤ 2.5 x ULN
* Estimated creatinine clearance of ≥ 40 mL/min using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) 2009 formula
* If not receiving anticoagulants: International normalized ratio (INR) OR prothrombin (PT) ≤ 1.5 x ULN
* If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants
* If not receiving anticoagulants: Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN
* If on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants
* Women of childbearing potential (WOCBP): Negative serum pregnancy test
* Agreement by females of childbearing potential to either abstain from heterosexual activity or use an effective method of birth control (failure rate of < 1% per year) during the treatment period and through at least 30 days after the last dose of venetoclax, 18 months after the last dose of obinutuzumab, 12 months after the last dose of epcoritamab, and at least 4 months after the last dose of tocilizumab (if applicable). Women must refrain from donating eggs during this same period

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)
  * Examples of contraceptive methods with a failure rate of < 1% per year include tubal ligation, male sterilization, hormonal implants, established, proper use of combined oral or injected hormonal contraceptives, and certain intrauterine devices
* Agreement by males to either abstain from heterosexual activity or use a condom during the treatment period and through at least 30 days after the last dose of venetoclax, 4 months after the last dose of obinutuzumab, epcoritamab or tocilizumab (as applicable). Men with a pregnant partner must agree to remain abstinent or use a condom for the duration of the pregnancy. Men must refrain from donating sperm during this same period

Exclusion Criteria:

* Chronic use of corticosteroids in excess of 20 mg/day prednisone or equivalent
* Major surgery (under general anesthesia) within 30 days prior to cycle 1 day 1 (C1D1)
* Uncontrolled coagulopathy or bleeding disorder. Direct oral anticoagulants are allowed
* Exposure to vaccination with live vaccine within 30 days prior to C1D1, or anticipated need for such vaccination during treatment
* Transformation of CLL to aggressive non-Hodgkin lymphoma (NHL) (Richter's transformation)
* Current evidence of central nervous system involvement by the CLL
* History of confirmed progressive multifocal leukoencephalopathy (PML)
* History of prior malignancy except:

  * Malignancy treated with curative intent and no known active disease present for ≥ 2 years prior to initiation of therapy on current study
  * Adequately treated non-melanoma skin cancer or lentigo maligna (melanoma in situ) without evidence of disease
  * Adequately treated in situ carcinomas (e.g., cervical, esophageal, etc.) without evidence of disease
  * Asymptomatic prostate cancer managed with "watch and wait" strategy
* Uncontrolled immune hemolysis or thrombocytopenia (positive direct antiglobulin test in absence of hemolysis or history of immune-mediated cytopenias are not exclusions)
* Uncontrolled active systemic infection
* Known positive test result for hepatitis C (hepatitis C virus [HCV] antibody serology testing) and a positive test result for HCV ribonucleic acid (RNA). Participants with positive serology are eligible in case of negative HCV RNA test results
* Known positive test result for chronic hepatitis B virus (HBV) infection (defined by hepatitis B virus surface antigen [HBsAg] positivity)

  * Participants with occult or prior HBV infection (defined as negative HBsAg and positive total hepatitis B core antibody) may be included if HBV deoxyribonucleic acid (DNA) is undetectable, provided that they are willing to undergo ongoing DNA testing
  * Antiviral prophylaxis may be administered as per institutional guidelines
  * Participants who have protective titers of hepatitis B virus surface antibody (HBsAb) after vaccination or prior but cured hepatitis B may be included if HBV DNA is undetectable
* Participants with HIV may be enrolled if they are on concurrent highly active antiretroviral therapy (HAART) therapy, have undetectable HIV RNA levels and no evidence of HIV-related comorbidities (infections or malignancies), and provided that they meet all other protocol-defined eligibility criteria
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2026-01-09 (Estimated); Primary Completion 2029-06-08 (Estimated); Study Completion 2029-06-08 (Estimated)

PRIMARY OUTCOMES:
Minimal residual disease (MRD) negative complete response (CR) | At beginning of cycle 12 (cycle length = 28 days)
  MRD status will be assessed using ClonoSEQ® (Adaptive Biotechnologies™) on the blood (sensitivity at 10^-4 and 10^-6). The determination of MRD status (i.e. positive versus negative) will be defined as the presence or absence of measurable clonotypes, respectively, at a sensitivity of 10^-6. Will be estimated along with the 95% exact binomial confidence interval.

SECONDARY OUTCOMES:
Overall response rate | After the start of protocol therapy and prior to disease progression and/or start of other anti-lymphoma therapy, assessed up to 5 years
  Will be defined as achieving a best response of either CR or partial response (PR) in a response-evaluable participant. Will be estimated along with the 95% exact binomial confidence interval.
Progression-free survival (PFS) | From start of protocol treatment to time of disease relapse/progression or death due to any cause, whichever occurs earlier, assessed up to 5 years
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval for survival at specific timepoints will be constructed based on log-log transformation. Median PFS will be estimated when possible.
Duration of response (DOR) | From the first achievement of PR or CR to time of disease relapse/progression or death, whichever earlier, assessed up to 5 years
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval for survival at specific timepoints will be constructed based on log-log transformation. Median DOR will be estimated when possible.
Overall survival (OS) | From start of protocol treatment to death due to any cause, assessed up to 5 years
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval for survival at specific timepoints will be constructed based on log-log transformation. Median OS will be estimated when possible.
Incidence of adverse events | Up to 60 days after last dose of study treatment
  Will be graded by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Hematologic toxicities will be graded according to International Workshop on Chronic Lymphocytic Leukemia. Cytokine release syndrome and immune effector cell associated neurotoxicity syndrome will be graded according to the American Society for Transplantation and Cellular Therapy Cytokine Release Syndrome Consensus Grading criteria. Observed toxicities will be summarized by type, severity, and attribution.

CONTACTS AND LOCATIONS:
Overall Officials: Alexey V Danilov, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (7):
- United States (7):
  - City of Hope Medical Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California
  - City of Hope at Long Beach Elm, Long Beach, California
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - City of Hope Atlanta Cancer Center, Newnan, Georgia
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Medical College of Wisconsin, Milwaukee, Wisconsin